CLINICAL TRIAL: NCT04546035
Title: Effect of Number of Pulses of Radial Extracorporeal Shock Wave Therapy on Hamstring Spasticity in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rizky Kusuma Wardhani (Other)
Responsible Party: Sponsor-Investigator, Rizky Kusuma Wardhani, M.D., Physiatrist, Consultant in PM&R Department, Indonesia University
Organization: Indonesia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LB.02/2.2/443/2020
Record Dates: First submitted 2020-08-24; First posted 2020-09-11 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Spasticity, Muscle; Cerebral Palsy; Child; Spastic
Keywords: Spasticity; Cerebral Palsy; Children; ESWT; Pulses
MeSH Terms: conditions — Muscle Spasticity; Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants (including parents of patients), physiatrists who conducted ESWT and physiatrists who examined the patients' ASAS score are all blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 500 pulses (Experimental): In this group, patients received one single rESWT session consisting of 500 pulses on hamstring muscle with energy flux density at 0.1 mJ/mm2, repetition frequency was at 4 Hz, and a pressure of 1.5 bars.
  Interventions: Device: radial Extracorporeal Shockwave Therapy
- 1,000 pulses (Experimental): In this group, patients received one single rESWT session consisting of 1,000 pulses on hamstring muscle with energy flux density at 0.1 mJ/mm2, repetition frequency was at 4 Hz, and a pressure of 1.5 bars.
  Interventions: Device: radial Extracorporeal Shockwave Therapy
- 1,500 pulses (Experimental): In this group, patients received one single rESWT session consisting of 1,500 pulses on hamstring muscle with energy flux density at 0.1 mJ/mm2, repetition frequency was at 4 Hz, and a pressure of 1.5 bars.
  Interventions: Device: radial Extracorporeal Shockwave Therapy
- 2,000 pulses (Experimental): In this group, patients received one single rESWT session consisting of 2,000 pulses on hamstring muscle with energy flux density at 0.1 mJ/mm2, repetition frequency was at 4 Hz, and a pressure of 1.5 bars.
  Interventions: Device: radial Extracorporeal Shockwave Therapy

INTERVENTIONS:
Device: radial Extracorporeal Shockwave Therapy — rESWT was given on hamstring muscles, with the subject lying on prone position. No anesthesia was required.
  Other Names: rESWT

SUMMARY:
Cerebral palsy (CP) is a group of permanent disorders affecting movement and postural development that are caused by non-progressive disruptions of the brain, usually occurring during fetal period or infancy. It is commonly accompanied with sensory disorders and learning disability. In 2016, more than 17 million people are affected by CP with a prevalence of 1.5 to 2.5 per 1,000 live births. CP remains to be the most common cause of severe physical disability in children. The Centres for Disease Control and Prevention (CDC) estimated an economic cost of US$4.1 million per CP patient that comprises of medical services, special education and productivity loss.

Current management of spasticity involves physical manipulation such as passive stretching and splinting, sometimes combined with oral pharmacologic treatment, intrathecal baclofen therapy and botulinum toxin injection. At times, surgical procedures such as Surgical Dorsal Rhizotomy (SDR) can also be considered. Botulinum toxin injection has been shown to reduce spasticity for up to 6 months, however, the cost of the procedure remains to be an issue in developing countries like Indonesia. Therefore, other modality such as a non-invasive therapy should be considered as an alternative treatment for spasticity.

Radial Extracorporeal Shockwave Therapy (rESWT) is a non-invasive treatment that has been shown to effectively improve spasticity in patients with spastic motor type CP, despite unclear underlying mechanism. According to International Society for Medical Shockwave Treatment (ISMST), there has yet to be a recommended guideline for the treatment of spasticity in children using rESWT. One crucial physical parameter needed to be determined is the number of pulse required to efficiently reduce spasticity. The number of pulse directly affects the duration of ESWT per session (the higher the number of pulse given, the longer the therapy session). This may be a concern for spastic motor type CP due to accompanying sensory and learning disability. Therefore, the objective of this study was to understand whether the reduction in hamstring stiffness in children with spastic CP could be influenced by the number of pulse in a single ESWT session.

DETAILED DESCRIPTION:
This study was designed as a double-blinded and randomized controlled trial.

Children with spastic CP from the outpatient clinic of the Department of Physical Medicine and Rehabilitation at Rumah Sakit Umum Pusat Nasional Dr. Cipto Mangunkusumo (RSCM) participated in the study. The patients were randomly allocated to four groups: 500 pulses, 1,000 pulses, 1,500 pulses, and 2,000 pulses. All groups undergo routine rehabilitation, including physiotherapy. Ethical approval was obtained from the Ethical Committee of Faculty of Medicine, University of Indonesia - RSCM.

Spasticity of hamstring was evaluated as the degree of resistance to passive movement using ASAS (0: no spasticity to 4: severe spasticity). Evaluations were done at four time points: 1) pre-ESWT, 2) immediately post-ESWT, 3) 2 weeks post-ESWT, and 4) 4 weeks post-ESWT. All patients were examined by the same physiatrist with the patient lying on supine position on the stretcher.

BTL-6000 SWT Topline (BTL, Czech Republic) was used to apply rESWT on hamstring muscles, with the subject lying on prone position. The energy flux density was constant at 0.1 mJ/mm2 and the repetition frequency was at 4 Hz, with a pressure of 1.5 bars. For double-blinded treatment, spastic hamstring muscles from CP patients were allocated into four groups - each group receiving a varying total number of pulses (group I: 500 pulses, group II: 1,000 pulses, group III: 1.500 pulses, and group IV: 2,000 pulses). No anesthesia was given. Adverse events were closely monitored during and after therapy.

Intra-group changes in ASAS were evaluated with Friedman analysis of variance from baseline immediately post ESWT, 2 weeks post ESWT, and 4 weeks post ESWT; followed by post-hoc Wilcoxon signed-ranked test. Inter-group differences in ASAS reduction were analyzed using Kruskal Wallis test. Statistical analysis was conducted using SPSS ver. 23.0 (IBM Corporation, Armonk, NY, USA). The level of significance was set at <0.05.

ELIGIBILITY:
Inclusion Criteria:

* patients with spastic CP aged 5 to 18 years old
* at least one hamstring with an Australian Spasticity Assessment Scale (ASAS) of 2 or more
* ability of legal respondent to give written informed consent

Exclusion Criteria:

* 6 months or less since the last botulinum injection on hamstring
* surgical operation on lower limb within the last 12 months
* severe contracture on hamstring

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-03-26 (Actual)

PRIMARY OUTCOMES:
Baseline Spasticity of Hamstring | Pre-ESWT
  Evaluated as the degree of resistance to passive movement using ASAS (0: no spasticity to 4: severe spasticity)
Spasticity of Hamstring immediately post-ESWT | Immediately post-ESWT
  Evaluated as the degree of resistance to passive movement using ASAS (0: no spasticity to 4: severe spasticity)
Spasticity of Hamstring 2 weeks post-ESWT | 2 weeks post-ESWT
  Evaluated as the degree of resistance to passive movement using ASAS (0: no spasticity to 4: severe spasticity)
Spasticity of Hamstring 4 weeks post-ESWT | 4 weeks post-ESWT
  Evaluated as the degree of resistance to passive movement using ASAS (0: no spasticity to 4: severe spasticity)

CONTACTS AND LOCATIONS:
Locations (1):
- Universitas Indonesia Fakultas Kedokteran, Jakarta Pusat, DKI Jakarta, Indonesia